CLINICAL TRIAL: NCT02847221
Title: Assessing Cough Peak Flow (CPF) Using Ventilator built-in Flow-meter to Predict Extubation Success: A Single Centre Study
Brief Title: Cough Peak Flow for Extubation Prediction
Acronym: CPF
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0495
Record Dates: First submitted 2016-07-25; First posted 2016-07-28 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Extubation in ICU Patients
Keywords: cough peak flow; scheduled weaning trial; scheduled extubation; prognosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Successful weaning from mechanical ventilation in ICU patients depends on patient ability to breathe spontaneously and on cough efficiency. Previous studies found that cough peak flow (CPF) at 60 L/min threshold predicted extubation failure. These studies measured CPF using a dedicated flow-meter that required patient disconnection from the ventilator, limiting the generalizability of this procedure. This study aimed to predict extubation outcome in a consecutive series of patients by measuring CPF from the ventilator flow-meter. CPF measurements were done by freezing ventilator screen and scrolling the cursor to the maximal value of CPF during expiration and Tidal Volume (TV) in preceding inspiration.

The objective was to assess the performance of CPF to predict early extubation outcome.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Intubation > 24h
* Eligible for scheduled weaning trial and then scheduled extubation
* Mechanical ventilation from Evita XL ventilator (Dräger, Germany)
* Patient's agreement to participate

Exclusion Criteria:

- Withdrawal decision of life supporting care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to a 15-bed medical ICU from November 1st 2014 to October 31st 2015
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2014-11; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Early extubation success rate (EES rate) | 48 hours
  Defining a relation between the CPF/TV ratio before extubation and early extubation success rate

SECONDARY OUTCOMES:
Scheduled weaning trial success rate | 48 hours
  Defining a relation between the CPF/TV ratio before weaning trial and scheduled weaning trial success rate

CONTACTS AND LOCATIONS:
Overall Officials: Florent GOBERT, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Medical Intensive care unit, Croix-Rousse Hospital. 103 Grande Rue de la Croix-Rousse, Lyon, France

REFERENCES:
- [Derived] Gobert F, Yonis H, Tapponnier R, Fernandez R, Labaune MA, Burle JF, Barbier J, Vincent B, Cleyet M, Richard JC, Guerin C. Predicting Extubation Outcome by Cough Peak Flow Measured Using a Built-in Ventilator Flow Meter. Respir Care. 2017 Dec;62(12):1505-1519. doi: 10.4187/respcare.05460. Epub 2017 Sep 12. PMID 28900041